CLINICAL TRIAL: NCT04485845
Title: Comparative Effecacy of Metformin and Vildagliptin on Cardiometabolic Risk Factors, Metabolic Syndrome, and Diabetic Nephropathy Progression
Brief Title: Metformin Versus Vildagliptin in Reducing Risk of Metabolic Syndrome Complications Progression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia K. Zaafar, lecturer of pharmacology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDE00218
Record Dates: First submitted 2020-03-24; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Metabolic Syndrome; Diabete Type 2; Kidney Insufficiency
Keywords: metfomin; vildagliptin; metabolic syndrome; T2DM; nephropathy
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Renal Insufficiency; Kidney Diseases | interventions — Vildagliptin; Captopril; Metformin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin treated group (Active Comparator): A group of patients treated with a daily dose of metformin
  Interventions: Drug: Captopril Tablets; Drug: MetFORMIN 500 Mg Oral Tablet
- vildagliptin treated group (Experimental): A group of patients treated with a daily dose of vildagliptin
  Interventions: Drug: Vildagliptin; Drug: Captopril Tablets

INTERVENTIONS:
Drug: Vildagliptin — to compare the effect of both metformin and vildagliptin on the progression of diabetes and metabolic complications and risk factors
  Arms: vildagliptin treated group
Drug: Captopril Tablets — used to treat hypertension in metabolic syndrome patients and as a renal protector
Drug: MetFORMIN 500 Mg Oral Tablet — antihyperglycemic drug for elevated plasma glucose level and help in weight loss for patients suffering from diabetes or metabolic syndrome
  Arms: metformin treated group

SUMMARY:
Several crosssectional and prospective studies have shown that metabolic syndrome and its related components are associated with both prevalent and incident CKD .

Although the mechanisms for these cardiovascular benefits of Metformin and vildagliptin remain unclear, they extend well beyond glycemic lowering, and therefore are probably best considered diverse "cardiometabolic" pharmaceuticals rather than simply type 2 diabetes drugs.

Metformin and vildagliptin have known vasculoprotective actions, but the value of these drugs on drug-naïve diabetic patients during 24 week use warrants investigation. The investigator's purpose was to observe their effects on weight control, Cardiometabolic Risk Factors, Metabolic Syndrome risk, and diabetic nephrooathy Progression.

DETAILED DESCRIPTION:
the current study is investigating the relation betweeneach componant of metabolic syndrome and kidney injury incidence or prevalence, and the mechanism of its occurence. the kidney protective effect of metformin and vildagliptin and the mechanism of this action whether it is related to their glucose lowering mechanism or not is also one of the important points to be investigated in the study

ELIGIBILITY:
Inclusion Criteria:

1. men or women 40-70 years of age
2. body mass index be-tween≥22 and ≤40 kg/m2.
3. DM with an HbA1c ≥ 7

Exclusion Criteria:

(1) pregnant or nursing women; (2) chronic (>7 consecutive days) oral, parenteral or intra-articular corticosteroid treatment within 8 weeks prior to Visit 1 (3) history or evidence of major hepatopathy (aspartate aminotransferase or alanineaminotransferase activities > 2.5 times the upper limit of normal) (4) ischemic heart disease or cerebrovascular disease (5) creatinine level > 0.133 mmol/L (6) major diabetes complications (chronic renal insufficiency, proliferative retinopathy and stroke); (7) extreme dyslipidemia, such as familial hypercholesterolaemia

-

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
progression of metabolic syndrome complications | 24 weeks
  investigate the effect of antidiabetic drugs on improving patients' cases and reduce complcations of metablic syndrome and that will be assessed by measuring glucose serum levels, insulin plasma levels to calculate insulin resistance by HOMA-ir
estimation of metabolic syndrome deterioration | 24 weeks
  study the effect of both antidiabetic drugs on blood pressure

SECONDARY OUTCOMES:
reduce nephropathic impairement | 24 weeks
  study the impact of both metformin and vildagliptin on reducing kidney deterioration for patients suffering from metabolic syndrome and that can be assessed by measuring kidney function serologically using ELISA kits for each parameter

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Zaafar, PhD, Principal Investigator — Lecturer of clinical pharmacology and toxicology
Locations (1):
- National Diabetes & Endocrinology Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No